CLINICAL TRIAL: NCT01584063
Title: Healthy Mothers on the Move
Acronym: Healthy MOMs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MOMS-2002
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2012-04

CONDITIONS: Pregnancy; Postpartum Period
Keywords: Mexican Americans; Pregnancy; Diabetes Mellitus Type 2; Prevention; Community health workers; Community based participatory research; Behavioral Intervention; Lifestyle Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): These women received general information about pregnancy and the postpartum period and tips for stress management. This information was delivered during 3 group meetings during pregnancy and 1 group meeting postpartum by trained staff from a local community mental health agency.
- MOMs Healthy Lifestyle Intervention (Experimental): These women received the culturally tailored Healthy MOMs Healthy Lifestyle Intervention, which included social support from Women's Health Advocates (community health workers) and peers, and the Healthy MOMs curriculum. This intervention curriculum covered topics related to healthy eating, physical activity, and stress management during pregnancy and postpartum. General information about pregnancy and the postpartum period were also provided. This intervention was delivered during 10 group meetings and 4 home visits.
  Interventions: Behavioral: Healthy MOMs Healthy Lifestyle Intervention

INTERVENTIONS:
Behavioral: Healthy MOMs Healthy Lifestyle Intervention — These women received the culturally tailored Healthy MOMs Healthy Lifestyle Intervention, which included social support from Women's Health Advocates (community health workers) and peers, and the Healthy MOMs curriculum. This intervention curriculum covered topics related to healthy eating, physical activity, and stress management during pregnancy and postpartum. General information about pregnancy and the postpartum period were also provided. This intervention was delivered during 10 group meetings and 4 home visits.
  Arms: MOMs Healthy Lifestyle Intervention

SUMMARY:
Healthy Mothers on the Move (Healthy MOMs), was a prospective randomized controlled trial that aimed to demonstrate the effectiveness of a healthy lifestyle intervention to reduce risk factors for obesity and type 2 diabetes. This behavioral intervention was tailored to the needs of pregnant and postpartum Latino women. This study was conducted between 2004 and 2006 in southwest Detroit.

DETAILED DESCRIPTION:
Specific Aims

1. Intervention group participants will have improved levels of protective behaviors (improved daily dietary composition and increased level of physical activity) that reduce the risk of type 2 diabetes compared to control group.
2. Intervention group participants will have improved their status on clinical measures of risk for type 2 diabetes (anthropometric and metabolic status) compared to the control group.
3. To assess whether theory-based variables, including changes in attitudes, behavioral and control beliefs, perceived social support and behavioral intention change from baseline, and whether these changes influence behavioral outcomes.
4. To identify aspects of project planning and implementation that contributed to achievement of behavioral and clinical outcomes. Measures include recruitment, retention and intervention participation rates, barriers and facilitators of participation; and community involvement in, and satisfaction with, intervention components and project activities; and fidelity of intervention components.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* A resident of Southwest Detroit
* Less than 20 weeks gestational at the eligibility screening

Exclusion Criteria: women with:

* Type 1 or type 2 diabetes
* Incompetent cervix/cerclage
* Active thyroid
* Multiple gestation
* Cardiac, vascular or pulmonary disease
* Drug or alcohol addiction
* Serious physical or mental illness or condition that would substantially interfere with participation in or completion of the entire intervention

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2004-02; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Diet
Physical Activity

SECONDARY OUTCOMES:
Weight (gain during pregnancy, postpartum retention)
Metabolic (e.g., glucose)

REFERENCES:
- [Derived] Shah MK, Kieffer EC, Choi H, Schumann C, Heisler M. Mediators and Moderators of the Effectiveness of a Community Health Worker Intervention That Improved Dietary Outcomes in Pregnant Latino Women. Health Educ Behav. 2015 Oct;42(5):593-603. doi: 10.1177/1090198114568307. Epub 2015 Jan 30. PMID 25636316
- [Derived] Kieffer EC, Welmerink DB, Sinco BR, Welch KB, Rees Clayton EM, Schumann CY, Uhley VE. Dietary outcomes in a Spanish-language randomized controlled diabetes prevention trial with pregnant Latinas. Am J Public Health. 2014 Mar;104(3):526-33. doi: 10.2105/AJPH.2012.301122. Epub 2013 Jun 13. PMID 23763411